CLINICAL TRIAL: NCT04371393
Title: Mesenchymal Stromal Cells for the Treatment of Moderate to Severe COVID-19 Acute Respiratory Distress Syndrome
Brief Title: MSCs in COVID-19 ARDS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: At 3d interim analysis, randomization, but not follow-up, was halted by the DSMB due to low predictive probability of achieving postulated mortality benefit (pre-specified 42.5% relative mortality reduction) were the trial to complete randomization.
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Mesoblast, Inc. (Industry); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Annetine Gelijns, Chair, Department of Population Health Science & Policy, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 08-1078-0014
Record Dates: First submitted 2020-04-28; First posted 2020-05-01 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Mesenchymal Stromal Cells; Remestemcel-L; Acute Respiratory Distress Syndrome; COVID
Keywords: mesenchymal stem cells; SARS-CoV-2; cytokine storm
MeSH Terms: conditions — Respiratory Distress Syndrome; Cytokine Release Syndrome | interventions — remestemcel-l

STUDY DESIGN:
Intervention Model Description: This will be a randomized (1:1 ratio), double blind, parallel design, placebo controlled trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This is a randomized clinical trial, in which the patients and investigators are masked to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Remestemcel-L Plus Standard of Care (Experimental): Intravenous infusion of remestemcel-L 2x10^6 MSC/kg of body weight plus standard of care
  Interventions: Biological: Remestemcel-L
- Placebo Plus Standard of Care (Placebo Comparator): Placebo (Plasma-Lyte) plus standard of care
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Remestemcel-L — administered twice during the first week, with the second infusion at 4 days following the first injection (± 1 day)
  Arms: Remestemcel-L Plus Standard of Care
Drug: Placebo — administered twice during the first week, with second infusion at 4 days following the first injection (± 1 day)
  Arms: Placebo Plus Standard of Care

SUMMARY:
The mortality rate in SARS-CoV-2-related severe ARDS is high despite treatment with antivirals, glucocorticoids, immunoglobulins, and ventilation. Preclinical and clinical evidence indicate that MSCs migrate to the lung and respond to the pro-inflammatory lung environment by releasing anti-inflammatory factors reducing the proliferation of pro-inflammatory cytokines while modulating regulatory T cells and macrophages to promote resolution of inflammation. Therefore, MSCs may have the potential to increase survival in management of COVID-19 induced ARDS.

The primary objective of this phase 3 trial is to evaluate the efficacy and safety of the addition of the mesenchymal stromal cell (MSC) remestemcel-L plus standard of care compared to placebo plus standard of care in patients with acute respiratory distress syndrome (ARDS) due to SARS-CoV-2. The secondary objective is to assess the impact of MSCs on inflammatory biomarkers.

DETAILED DESCRIPTION:
This will be a randomized (1:1 ratio), double blind, parallel design, placebo controlled trial. Randomization will be stratified by clinical center and by moderate versus severe ARDS. The study is designed to have three interim analyses for stopping accrual early for efficacy and futility when 30%, 45% and 60% of the 300 patients have reached the primary endpoint using Bayesian predictive probabilities.

Patients will be randomized in a 1:1 allocation to intravenous infusion of MSCs (remestemcel-L) plus standard of care versus placebo plus standard of care for the treatment of COVID-19 related ARDS:

* Group 1: 2x10^6 MSC/kg of body weight plus standard of care, administered twice during the first week, with the second infusion at 4 days following the first infusion (± 1 day)
* Group 2: Placebo (Plasma-Lyte) plus standard of care, administered twice during the first week, with the second infusion at 4 days following the first infusion (± 1 day) (control)

MSCs and placebo will initially be administered intravenously in the dose defined above at randomization. The rate of infusion may be tailored to the patient's respiratory status and fluid status, but the duration of infusion should not exceed 60 minutes.

Patients will be followed for 90 days post randomization, with assessment of pulmonary symptoms at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria

* 18 years or older
* Patient has SARS-CoV-2 (COVID-19) confirmed by real-time reverse transcription polymerase chain reaction (RT-PCR) assay or other diagnostic test
* Patient requiring mechanical ventilatory support with moderate to severe ARDS as determined by the following criteria (adapted from the Berlin criteria)

  * Bilateral opacities must be present on a chest radiograph or computerized tomographic (CT) scan. These opacities are not fully explained by pleural effusions, lobar collapse, lung collapse, or pulmonary nodules.
  * Respiratory failure not fully explained by cardiac failure or fluid overload.
  * Moderate to severe impairment of oxygenation must be present, as defined by the ratio of arterial oxygen tension to fraction of inspired oxygen (PaO2/FiO2). The severity of the hypoxemia defines the severity of the ARDS:
* Moderate ARDS: PaO2/FiO2 >100 mmHg and ≤200 mmHg, on ventilator settings that include PEEP ≥5 cm H2O OR
* Severe ARDS: PaO2/FiO2 ≤100 mmHg on ventilator settings that include PEEP ≥5 cm H2O
* High sensitivity C-Reactive Protein (hs-CRP) or CRP serum level >4.0 mg/dL
* Acute Physiologic and Chronic Health Evaluation (APACHE IV) score >5
* Creatinine clearance of ≥ 30 mL/minute OR a creatinine clearance of 20-29 mL/minute with urine output of ≥0.3 mLs/kg/hour over the last 8 hours or ≥500 mLs over the last 24 hours
* The patient or his/her legally authorized representative (LAR) is able to provide informed consent

Exclusion Criteria

* Currently receiving extracorporeal membrane oxygenation (ECMO) or high frequency oscillatory ventilation (HFOV)
* Females who are pregnant or lactating
* Patients with established positive bacterial blood cultures prior to enrollment or suspicion of superimposed bacterial pneumonia
* Patients with BMI >55
* Patients with untreated HIV infection
* Patients with malignancy who are within 12 months of active treatment with any chemotherapy, radiation or immunotherapy.
* Patients who have been intubated for more than 72 hours in total at the time of randomization
* Creatinine clearance less than 20 mL/minute or receiving renal replacement therapy
* LFTs (isolated ALT or AST) > 8x upper limit of normal or > 5x upper limit of normal in the setting of other liver function abnormalities (i.e., total bilirubin ≥ 2x upper limit of normal)
* Known hypersensitivity to DMSO or to porcine or bovine proteins
* History of prior respiratory disease with requirement for supplemental oxygen
* Any end-stage organ disease which in the opinion of the investigator may possibly affect the safety of remestemcel-L treatment
* Receiving an investigational cellular therapy agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2022-01-02 (Actual)

PRIMARY OUTCOMES:
Number of all-cause mortality | 30 days
  Number of all-cause mortality within 30 days of randomization.

SECONDARY OUTCOMES:
Number of days alive off mechanical ventilatory support | 60 days
  Number of days alive off mechanical ventilatory support calculated as the number of days, within the 60 days window, that patients were alive and free of mechanical ventilatory support.
Number of adverse events | 30 days
  Safety analyses will be assessed by adverse event rates calculated as the ratio of the total number of events over 30 days divided by total patient-time at risk for the specific event from randomization.
Number of participants alive at day 7 | 7 days
Number of participants alive at day 14 | 14 days
Number of participants alive at day 60 | 60 days
Number of participants alive at day 90 | 90 days
Number of participants alive at 12 Months | 12 Months
Number of participants with resolution and/or improvement of ARDS | 7 days
  The number and percent of patients with resolution and/or improvement of ARDS at day 7
Number of participants with resolution and/or improvement of ARDS | 14 days
  The number and percent of patients with resolution and/or improvement of ARDS at day 14
Number of participants with resolution and/or improvement of ARDS | 21 days
  The number and percent of patients with resolution and/or improvement of ARDS at day 21
Number of participants with resolution and/or improvement of ARDS | 30 days
  The number and percent of patients with resolution and/or improvement of ARDS at day 30
Severity of ARDS | baseline and 7 days
  severity of ARDS according to Berlin Criteria at days 7 post-randomization Change from baseline of the severity of ARDS according to Berlin Criteria at days 7, 14, 21 and 30 post-randomization will be compared between treatment groups using a Cochran-Mantel-Haenszel test stratified by baseline severity.
Severity of ARDS | baseline and 14 days
  severity of ARDS according to Berlin Criteria at days 14 post-randomization Change from baseline of the severity of ARDS according to Berlin Criteria at days 7, 14, 21 and 30 post-randomization will be compared between treatment groups using a Cochran-Mantel-Haenszel test stratified by baseline severity.
Severity of ARDS | baseline and 21 days
  severity of ARDS according to Berlin Criteria at days 21 post-randomization Change from baseline of the severity of ARDS according to Berlin Criteria at days 7, 14, 21 and 30 post-randomization will be compared between treatment groups using a Cochran-Mantel-Haenszel test stratified by baseline severity.
Severity of ARDS | baseline and 30 days
  severity of ARDS according to Berlin Criteria at days 30 post-randomization Change from baseline of the severity of ARDS according to Berlin Criteria at days 7, 14, 21 and 30 post-randomization will be compared between treatment groups using a Cochran-Mantel-Haenszel test stratified by baseline severity.
Length of stay | 12 months
  Hospital length of stay
Readmissions | 12 months
  number of readmission
Length of Stay in Intensive Care Unit | 12 months
Clinical Improvement Scale | 7 days
  Change from baseline in Clinical Improvement Scale at day 7. Clinical Improvement Scale full scale from 1 to 7, with higher score indicating more clinical improvement.
Clinical Improvement Scale | 14 days
  Change from baseline in Clinical Improvement Scale at day 14. Full scale from 1 to 7, with higher score indicating more clinical improvement.
Clinical Improvement Scale | 21 days
  Change from baseline in Clinical Improvement Scale at day 21. Clinical Improvement Scale full scale from 1 to 7, with higher score indicating more clinical improvement.
Clinical Improvement Scale | 30 days
  Change from baseline in Clinical Improvement Scale at day 30. Clinical Improvement Scale full scale from 1 to 7, with higher score indicating more clinical improvement.
Change in plasma hs-CRP concentration | baseline and 7 days
  Changes from baseline in plasma hs-CRP concentration at days 7
Change in plasma hs-CRP concentration | baseline and 14 days
  Changes from baseline in plasma hs-CRP concentration at days 14
Change in plasma hs-CRP concentration | baseline and 21 days
  Changes from baseline in plasma hs-CRP concentration at days 21
Change in serum hs-CRP concentration | baseline and 30 days
  Changes from baseline in serum hs-CRP concentration at days 30
Change in IL-6 inflammatory marker level | baseline and 7 days
  Changes from baseline in IL-6 inflammatory marker level at 7 days
Change in IL-6 inflammatory marker level | baseline and 14 days
  Changes from baseline in IL-6 inflammatory marker level at 14 days
Change in IL-6 inflammatory marker level | baseline and 21 days
  Changes from baseline in IL-6 inflammatory marker level at 21 days
Change in IL-6 inflammatory marker level | baseline and 30 days
  Changes from baseline in IL-6 inflammatory marker level at 30 days
Change in IL-8 inflammatory marker level | baseline and 7 days
  Changes from baseline in IL-6 inflammatory marker level at 7 days
Change in IL-8 inflammatory marker level | baseline and 21 days
  Changes from baseline in IL-6 inflammatory marker level at 21 days
Change in IL-8 inflammatory marker level | baseline and 14 days
  Changes from baseline in IL-6 inflammatory marker level at 14 days
Change in IL-8 inflammatory marker level | baseline and 30 days
  Changes from baseline in IL-6 inflammatory marker level at 30 days
Change in TNF-alpha inflammatory marker level | baseline and 7 days
  Changes from baseline in TNF-alpha inflammatory marker level at 7 days
Change in TNF-alpha inflammatory marker level | baseline and 14 days
  Changes from baseline in TNF-alpha inflammatory marker level at 14 days
Change in TNF-alpha inflammatory marker level | baseline and 21 days
  Changes from baseline in TNF-alpha inflammatory marker level at 21 days
Change in TNF-alpha inflammatory marker level | baseline and 30 days
  Changes from baseline in TNF-alpha inflammatory marker level at 30 days
Pulmonary symptoms | 6 months
  including the presence of emphysema, COPD, asthma, pulmonary fibrosis, other pulmonary disease, and the need for respiratory support will be reported by randomization
Pulmonary symptoms | 12 months
  including the presence of emphysema, COPD, asthma, pulmonary fibrosis, other pulmonary disease, and the need for respiratory support will be reported by randomization

CONTACTS AND LOCATIONS:
Overall Officials: Annetine C Gelijns, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Michael Mack, MD, Study Director — Baylor Research Institute; Peter Smith, MD, Study Director — Duke University
Locations (21):
- United States (21):
  - Dignity Health, Gilbert, Arizona
  - University of Southern California, Los Angeles, California
  - Stanford University, Stanford, California
  - Emory University, Atlanta, Georgia
  - Lutheran Hospital, Fort Wayne, Indiana
  - Ochsner Clinic, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - University of Maryland, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Dartmouth-Hitchcock, Lebanon, New Hampshire
  - New York University Langone Health, New York, New York
  - Mount Sinai Health, New York, New York
  - Northwell Health, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - WakeMed, Raleigh, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Houston Methodist Hospital, Houston, Texas
  - Baylor, Smith & White, Plano, Texas
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: De-identified study data sets must be submitted to the designated NHLBI Program Official no later than 3 years after the end of the clinical activity (final patient follow-up, etc.) or 2 years after the main paper of the trial has been published, whichever comes first. Data are prepared by the study coordinating center and sent to the designated PO for review prior to release.
Access Criteria: Anyone who wishes to access the data.